CLINICAL TRIAL: NCT06205641
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study on the Efficacy and Safety of Xuanfei Baidu Granule in the Treatment of Influenza A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Zhaohui Tong, Derictor of Beijing Institute of Respiratory Diseases and Vice president of Beijing Chaoyang Hospital, Capital Medical University, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XFBD-JL-001
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Influenza A
Keywords: Influenza A; Xuanfei Baidu Granule
MeSH Terms: interventions — baloxavir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Xuanfei Baidu Granule Placebo group (Placebo Comparator)
  Interventions: Drug: Xuanfei Baidu Granule Placebo
- Xuanfei Baidu Granule group (Experimental)
  Interventions: Drug: Xuanfei Baidu Granule
- Baloxavir Marboxil Tablet group (Active Comparator)
  Interventions: Drug: Baloxavir Marboxil Tablet
- Combination group (Active Comparator)
  Interventions: Drug: Xuanfei Baidu Granule; Drug: Baloxavir Marboxil Tablet

INTERVENTIONS:
Drug: Xuanfei Baidu Granule Placebo — Take Xuanfei Baidu Granule Placebo 1 bag in the morning and evening with boiling water for 5 days.
  Arms: Xuanfei Baidu Granule Placebo group
Drug: Xuanfei Baidu Granule — Take Xuanfei Baidu Granule 1 bag in the morning and evening with boiling water for 5 days.
  Arms: Combination group; Xuanfei Baidu Granule group
Drug: Baloxavir Marboxil Tablet — Take Baloxavir Marboxil Tablet 2 tablets orally, once a day, for 1 day.
  Arms: Baloxavir Marboxil Tablet group; Combination group

SUMMARY:
This study is a prospective, multicenter, randomized controlled trial and aims to evaluate efficacy and safety of Xuanfei Baidu Granule in the treatment of influenza A.

This study plans to enroll 584 subjects. The subjects will be randomly divided into 4 groups according to the ratio of 1:1:1:1, and they will be treated with Xuanfei Baidu Granule Placebo, Xuanfei Baidu Granule, Xuanfei Baidu Granule combined with Baloxavir Marboxil tablet.1 bag of Xuanfei Baidu Granule and Xuanfei Baidu Granule Placebo in the morning and evening, and take with boiling water for 5 days. Baloxavir Marboxil Tablet was taken orally 2 tablets, once a day for 1 day.

The subjects were visited every day for 7 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥18 and <65, regardless of gender.
* Meet the western medicine diagnostic criteria for influenza in the "2020 Edition of the Diagnosis and Treatment Scheme for Influenza".
* Onset of illness within ≤72 hour.
* Body temperature ≥37.5℃ within 24 hours before treatment.
* Tested positive for influenza A virus by antigen.
* The subject understands and voluntarily signs the informed consent, and is able to follow the visit and related procedures prescribed by the program.

Exclusion Criteria:

* Individuals with known allergies to the test drugs, placebo components, or having allergic constitution.
* Meet the criteria for severe or critical cases as per the "2020 Edition of the Diagnosis and Treatment Scheme for Influenza".
* Patients with acute bacterial sinusitis, allergic rhinitis, tracheitis-bronchitis, pneumonia, herpetic pharyngitis, or similar diseases.
* Individuals with severe primary diseases in cardiovascular, pulmonary, hepatic, renal, and hematopoietic systems.
* Patients with mental illness or those unable or unwilling to cooperate.
* History of epilepsy or febrile convulsions.
* Obesity (BMI >30).
* Patients with acute and chronic gastroenteritis and unexplained diarrhea within 1 week before administration.
* Liver function test values (ALT, AST) exceed 60U/L;Serum creatinine over 106μmol/L.
* Use of other drugs for the treatment of the disease within 24 hours before administration (including antiviral, hormone and other Chinese and Western drugs and treatment methods).
* Suspected or confirmed history of alcohol or drug abuse, heavy smoker.
* Women who are pregnant or trying to become pregnant, breastfeeding women, those of childbearing age who are unable or unwilling to use adequate contraception during the trial or whose spouse is unwilling to use contraception.
* Immunodeficient, immunosuppressed patients or those who have received steroid therapy or other immunosuppressive therapy in the last 3 months.
* Received influenza vaccine within the last 12 months.
* Participants who have participated in other interventional clinical trials within the last 3 months.
* Participants considered unsuitable for this clinical trial by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The time to fever resolution. | within 7 days of enrollment
  Definition of fever resolution: the body temperature drops to ≤37 ℃ and is maintained for more than 24 hours.
  Definition of time to fever resolution: the time from the first dose to the resolution of fever.

SECONDARY OUTCOMES:
The time to alleviation of influenza symptoms. | within 7 days of enrollment
  Influenza symptoms include cough, sore throat, headache, stuffy nose, chills/sweating (feeling hot), muscle aches and fatigue.
  Influenza symptoms was measured by Influenza Symptom Rating Scale.The minimum and maximum value of every symptom is 0 and 3, respectively. Higher score means a worse outcome.
  Definition of alleviation of influenza symptoms: symptom score ≤1. Definition of time to alleviation of influenza symptoms: the time from the first dose to symptom improvement.
The proportion of patients with fever resolution. | within 7 days of enrollment
  Definition of fever resolution: the body temperature drops to ≤37 ℃ and is maintained for more than 24 hours.
The proportion of patients with alleviation of influenza symptoms. | within 7 days of enrollment
  Influenza symptoms include cough, sore throat, headache, stuffy nose, chills/sweating (feeling hot), muscle aches and fatigue.
  Influenza symptoms was measured by Influenza Symptom Rating Scale.The minimum and maximum value of every symptom is 0 and 3, respectively. Higher score means a worse outcome.
  Definition of alleviation of influenza symptoms: symptom score ≤1.
The proportion of patients with alleviation of clinical symptoms. | within 7 days of enrollment
  Clinical symptoms include fever resolution and alleviation of influenza symptoms.
  Influenza symptoms include cough, sore throat, headache, stuffy nose, chills/sweating (feeling hot), muscle aches and fatigue.
  Influenza symptoms was measured by Influenza Symptom Rating Scale.The minimum and maximum value of every symptom is 0 and 3, respectively. Higher score means a worse outcome.
  Definition of fever resolution: the body temperature drops to ≤37 ℃ and is maintained for more than 24 hours.
  Definition of alleviation of influenza symptoms: symptom score ≤1.
The temporal variation of body temperature. | within 7 days of enrollment
  The temperature was measured at 8 o 'clock, 12 o 'clock, 16 o 'clock and 20 o 'clock every day, and the measurement time and measurement results were recorded.
The temporal variation of Influenza Symptom Rating Scale. | within 7 days of enrollment
  Influenza symptoms include cough, sore throat, headache, stuffy nose, chills/sweating (feeling hot), muscle aches and fatigue.
  Influenza symptoms was measured by Influenza Symptom Rating Scale.The minimum and maximum value of every symptom is 0 and 3, respectively. Higher score means a worse outcome.
All-cause hospitalization rate. | within 7 days of enrollment
  All-cause hospitalization rate.
The incidence of clinical abnormalities was examined in the laboratory. | within 7 days of enrollment
  The incidence of clinical abnormalities was examined in the laboratory.
The incidence of clinical abnormalities was examined by electrocardiogram. | within 7 days of enrollment
  The incidence of clinical abnormalities was examined by electrocardiogram.
The incidence of all-cause adverse events during the study period. | within 7 days of enrollment
  The incidence of all-cause adverse events during the study period.
The incidence of serious adverse events during the study period. | within 7 days of enrollment
  The incidence of serious adverse events during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No